CLINICAL TRIAL: NCT05496608
Title: Treatment of Periodontal Intrabony Defects With Dense Leukocyte and Platelet-Rich Fibrin (L-PRF) Membrane Alone or in Combination With Collagen Membranes (Randomized Clinical and Biochemical Trial)
Brief Title: Treatment of Intrabony Defects With L-PRF Membrane With or Without Collagen Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Ramy Mubarak Hussein, Principal investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ainshams University
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Periodontal Bone Loss; Periodontal Diseases
MeSH Terms: conditions — Alveolar Bone Loss; Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: * The clinical data (Gingival index, Plaque index, PPD, CAL) were collected by a blinded single operator at the university outpatient clinic.
  * The biochemical analysis: The biochemist received the filter papers with a label for group letter and patient number. She was didn't know which intervention was carried out for any of the samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open Flap Debridement (Placebo Comparator): Subjects with infrabony defects had full thickness flap reflection and debridement of periodontal lesion
  Interventions: Procedure: OFD
- L-PRF (Active Comparator): Subjects with infrabony defects had full thickness flap reflection and debridement of periodontal lesion followed by application of the L-PRF within the bony defect
  Interventions: Procedure: L-PRF; Procedure: OFD
- L-PRF + CM (Active Comparator): Subjects with infrabony defects had full thickness flap reflection and debridement of periodontal lesion followed by application of the L-PRF within the bony defect and coverage with collagen xenogeneic membrane
  Interventions: Procedure: L-PRF; Procedure: OFD; Procedure: CM

INTERVENTIONS:
Procedure: L-PRF — a blood sample is obtained from the patient, and centrifuged to prepare a leukocyte platelet rich fibrin harvest that is applied within the derided lesion.
  Other Names: Leukocyte platelet rich fibrin
  Arms: L-PRF; L-PRF + CM
Procedure: OFD — Full thickness flap elevation to gain access to the infrabony lesion for debridement followed by flap closure.
  Other Names: Open flap Debridement
Procedure: CM — Xenogeneic collagen membranes that are used as barrier membranes in guided tissue regeneration of periodontal defects
  Other Names: Collagen membrane
  Arms: L-PRF + CM

SUMMARY:
For patients having periodontal intrabony lesions, three treatment modalities were executed to evaluate the effect of protecting Leukocyte rich -Platelet Rich Fibrin harvests (applied in the bony defects) with resorbable collagen membranes. Clinical Outcomes recorded were the Plaque index (PI), Gingival index (GI), probing depth reduction (PD), Clinical attachment level (CAL), and radiographic defect depth changes.

For the biochemical evaluation: levels of PDGF-BB and VEGF obtained from crevicular fluid by Perio-Paper strips were assessed using ELIZA.

DETAILED DESCRIPTION:
* Patients having 2-3 osseous bony wall infrabony periodontal lesions are enrolled in the present study. They have to be free from any systemic disease that contraindicates periodontal surgeries.
* Baseline data are obtained including the GI, PI, PD, CAL and preoperative paralleling periapical radiographs.
* Full thickness mucoperiosteal flaps are elevated and thorough debridement of the periodontal bony defect is performed.
* for OFD group; following debridement and saline irrigation, wound closure proceeds.
* for the L-PRF group; L-PRF is prepared and applied within the defect before primary closure.
* for the L-PRF + CM: similar procedure like the second group is performed but with an additional protective layer of collagen membrane on top of the defect before wound closure.
* from the second day postoperative; Periopaper strips are used to obtain a crevicular fluid sample from the sulcus
* At 6 months postoperative: the same baseline clinical measurements are obtained.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of one interproximal pocket probing depth of ≥6 mm and/or ≥5 mm CAL after 4 weeks from phase I execution
* 2 or 3 osseous wall interproximal intrabony defects that are ≥3mm in depth

Exclusion Criteria:

* Systemic diseases or conditions that contraindicate periodontal surgeries and/or affect the formed elements of the blood
* Patients who received antibiotic therapy and/or anti-inflammatory drug within the past 6 months
* Vulnerable groups
* Interdental craters and 1 wall osseous defects
* Active periapical pathosis

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Gingival index | 6 months
  measures the score of gingival inflammation. Minimum value of 0: denotes absence of inflammation. Maximum value = 3 and denotes severe inflammation
Plaque index | 6 months
  measures the score of plaque accumulation. Minimum value of 0: denotes absence of plaque on teeth surfaces. Maximum value = 3 and denotes diffuse and abundant plaque accumulation on teeth surfaces
Probing depth | 6 months
  measures the reduction in pocket depth
Clinical attachment level | 6 months
  measures the changes in amount of periodontal attachment
CEJ to base of defect | 6 months
  measures the changes in bone defect depth
CEJ to alveolar crest | 6 months
  measures the amount of crystal bone changes

SECONDARY OUTCOMES:
PDGF | 31 days
  Biochemical Evaluation of changes in levels of crevicular Platelet Derived Growth Factor -BB
VEGF | 31 days
  Biochemical Evaluation of changes in levels of crevicular Vascular endothelial growth factor

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gamal, P.H.D, Study Chair — Professor of periodontology
Locations (1):
- Ainshams University, Cairo, Egypt

REFERENCES:
- [Derived] Mubarak R, Adel-Khattab D, Abdel-Ghaffar KA, Gamal AY. Adjunctive effect of collagen membrane coverage to L-PRF in the treatment of periodontal intrabony defects: a randomized controlled clinical trial with biochemical assessment. BMC Oral Health. 2023 Sep 4;23(1):631. doi: 10.1186/s12903-023-03332-0. PMID 37667213